CLINICAL TRIAL: NCT00354744
Title: Intensive Multi-Agent Therapy, Including Dose-Compressed Cycles of Ifosfamide/Etoposide (IE) and Vincristine/Doxorubicin/Cyclophosphamide (VDC) for Patients With High-Risk Rhabdomyosarcoma
Brief Title: High-Dose Combination Chemotherapy and Radiation Therapy in Treating Patients With Newly Diagnosed Metastatic Rhabdomyosarcoma or Ectomesenchymoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARST0431; CDR0000489215 (Other: Clinical Trials.gov); COG-ARST0431 (Other: Children's Oncology Group)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2019-02

CONDITIONS: Sarcoma
Keywords: adult rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; adult malignant mesenchymoma; childhood malignant mesenchymoma; metastatic childhood soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Rhabdomyosarcoma; Malignant mesenchymal tumor | interventions — Dactinomycin; Cyclophosphamide; Doxorubicin; Etoposide; etoposide phosphate; Ifosfamide; Irinotecan; Vincristine; Radiotherapy; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Risk Rhabdomyosarcoma (Experimental): Parameningeal (without intracranial extension) and paraspinal tumors receive chemotherapy starting Week 1 and begin radiation therapy at Week 20. Weeks 1-6: vincristine sulfate and irinotecan hydrochloride. Weeks 7-34: vincristine sulfate and irinotecan hydrochloride, Cyclophosphamide with MESNA, Doxorubicin hydrochloride, Etoposide, Ifosfamide with MESNA. Weeks 35-54: vincristine sulfate, Dactinomycin, irinotecan hydrochloride and Cyclophosphamide with MESNA and Filgrastim. Radiation therapy beginning at Week 20. Second look conventional surgery: Surgical resection other than biopsy will be applicable for the majority of patients.
  Interventions: Biological: dactinomycin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Drug: irinotecan hydrochloride; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy; Biological: filgrastim

INTERVENTIONS:
Biological: dactinomycin — Age based dosage: ≥ 1 year 0.045 mg/kg IV x 1(maximum dose 2.5 mg), < 1 year 0.025 mg/kg.
  Day 1 of Weeks 35, 38, 41 and 44.
  Given IV
  Other Names: Actinomycin-D; Cosmegen; NSC #3053
Drug: cyclophosphamide — Age based dosage: ≥ 3 years 1200 mg/m2, <3 years 40 mg/kg.
  Day 1 of weeks 7, 11, 15, 28, 32, 35, 38, 41 and 44.
  Given IV
  Other Names: Cytoxan; NSC #26271
Drug: doxorubicin hydrochloride — Age based dosage: ≥ 1 year: 37.5mg/m²/day, < 1 year: treat with 50% doses calculated on a m2 basis. Total dose 75 mg/m².
  Days 1 and 2 of weeks 7, 11, 15, 28 and 32.
  Given IV
  Other Names: Adriamycin; NSC #123127
Drug: etoposide — Age based dosage: ≥ 1 year: 100 mg/m²/day, < 1 year: treat with 50% doses calculated on a m2 basis.
  Days 1-5 of weeks 9, 13, 17, 26 and 30.
  Given IV
  Other Names: VePesid; Etopophos; VP-16; NSC #141540
Drug: ifosfamide — Age based dosage: ≥ 1 year: 1800 mg/m²/day, < 1 year: treat with 50% doses calculated on a m2 basis.
  Days 1-5 of weeks 9, 13, 17, 26 and 30.
  Given IV
  Other Names: Isophosphamide; Iphosphamide; Z4942; Ifex; NSC #109724
Drug: irinotecan hydrochloride — Dosage 50 mg/m2-max dose 100 mg/day.
  Days 1-5 of weeks 1, 4, 20, 23, 47 and 50.
  Given IV
  Other Names: CPT-11; Camptothecin-11; 7-ethyl-10-(4-[1-piperidino]-1-piperidino)-carbonyloxy-camptothecin; Camptosar; NSC #616348
Drug: vincristine sulfate — Age based dosage: ≥ 3 years 1.5 mg/m2 (max dose 2 mg), ≥ 1 year and < 3 years 0.05 mg/kg (max dose 2 mg), < 1 year 0.025 mg/kg.
  Days 1-5 of weeks 1, 2, 3, 4, 5, 7, 8, 11, 12, 15, 16, 20, 21, 22, 23, 24, 28, 29, 32, 33, 35, 38, 41, 42, 43, 44, 47, 48, 50, and 51.
  Given IV
  Other Names: Oncovin; VCR; LCR; NSC #67574
Procedure: conventional surgery — Resection of the primary tumor with a surrounding "envelope" of normal tissue
Radiation: radiation therapy — Radiotherapy beginning at Week 20 to the primary tumor and to the metastatic sites excepting those with parameningeal tumors with intracranial extension (direct extension into the brain) and those requiring emergency radiotherapy
Biological: filgrastim — 5 micrograms/kg/day (max 300 micrograms) beginning 24-36 hours after the last dose of chemotherapy. Continue at least 7 days, or until the ANC ≥750/μL whichever comes last.
  Given subcutaneously.
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vincristine, irinotecan, ifosfamide, etoposide, doxorubicin, cyclophosphamide, and dactinomycin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving high-dose combination chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase III trial is studying how well giving high-dose combination chemotherapy together with radiation therapy works in treating patients with newly diagnosed metastatic rhabdomyosarcoma or ectomesenchymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Improve the early disease control interval for patients with newly diagnosed, high-risk, metastatic rhabdomyosarcoma or ectomesenchymoma using intensive, interval-compression therapy (comprising vincristine, irinotecan hydrochloride, ifosfamide, etoposide, doxorubicin hydrochloride, cyclophosphamide, and dactinomycin) that permits maximal early exposure to known effective agents.
* Determine the feasibility and assess immediate- and short-term side effects of concurrent irinotecan hydrochloride and radiotherapy in these patients.

Secondary

* Expand the available data for response to irinotecan hydrochloride and vincristine in previously untreated patients with high-risk rhabdomyosarcoma.
* Evaluate, prospectively, and validate gene expression values with the intent to define the best diagnostic predictors and more powerful prognostic classifiers.

OUTLINE: This is a prospective, nonrandomized, multicenter study. Patients are stratified according to prognostic factors predictive of outcome (e.g. histology, bone/bone marrow involvement, and number of metastatic sites).

Patients receive high-dose chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-5, 7, 8, 11, 12, 15, 16, 20-24, 28, 29, 32, 33, 35, 38, 41-44, 47, 48, 50, and 51; irinotecan hydrochloride IV over 1 hour on days 1-5 of weeks 1, 4, 20, 23, 47, and 50; and ifosfamide IV over 1 hour and etoposide IV over 30-60 minutes on days 1-5 of weeks 9, 13, 17, 26, and 30. Patients also receive doxorubicin hydrochloride IV continuously over 24 hours on days 1 and 2 of weeks 7*, 11, 15, 28, and 32; cyclophosphamide IV over 30-60 minutes on day 1 of weeks 7, 11, 15, 28, 32, 35, 38, 41, and 44; and dactinomycin IV over 1-5 minutes on day 1 of weeks 35, 38, 41, and 44 in the absence of disease progression or unacceptable toxicity. Patients also receive filgrastim (G-CSF) subcutaneously in weeks 7-9, 11-13, 15-17, 22, 26, 28-30, 32, 33, 35, 38, and 41-44 beginning 24-36 hours after the last chemotherapy dose and continuing until blood counts recover.

NOTE: *Patients undergoing early radiotherapy for intracranial extension do not receive doxorubicin in week 7.

Beginning at week 20 (or week 1 for patients with parameningeal tumors with intracranial extension [or spinal cord compression] requiring emergency radiotherapy), patients also undergo radiotherapy once a day, 5 days a week, for approximately 5½ weeks. Some patients may also undergo second-look surgery.

After completion of study treatment, patients are followed periodically for ≥ 10 years.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed high-risk rhabdomyosarcoma or ectomesenchymoma

  * Prior enrollment on COG-D9902 to confirm local histological diagnosis required

    * Tissue must be submitted for pathologic review within 2 days of patient registration on COG-D9902
  * Newly diagnosed disease
  * Metastatic disease (stage IV, clinical group IV)
* Has undergone initial surgical procedure (including biopsy) that provided the definitive diagnosis within the past 42 days
* Parameningeal and paraspinal tumors allowed

  * Patients with parameningeal (without intracranial extension [ICE]) and paraspinal tumors should begin study chemotherapy at week 1 and radiotherapy at week 20
* Patients with evidence of ICE, as defined by contrast MRI showing that primary tumor touches, displaces, invades, distorts, or otherwise causes a signal abnormality of the dura in contiguity to the primary site in brain or spinal cord, are eligible

  * ICE is presumed to exist if the cerebrospinal fluid cytopathology is positive for tumor at diagnosis
* Patients requiring emergency radiotherapy are eligible

  * Patients requiring emergency radiotherapy (for intracranial extension or spinal cord impingement) should begin study chemotherapy at week 1 (irinotecan hydrochloride and vincristine) concurrently with radiation therapy

PATIENT CHARACTERISTICS:

* ECOG or Zubrod performance status (PS) 0-2 (Lansky PS 50-100% for patients < 10 years of age and Karnofsky PS 50-100% for patients ≥ 10 years of age)
* Absolute neutrophil count ≥ 750/mm³*
* Platelet count ≥ 75,000/mm³*
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min (≥ 40 mL/min for infants < 1 year of age)
* Patients with urinary tract obstruction by tumor must meet the renal function criteria listed above AND must have unimpeded urinary flow established via decompression of the obstructed portion of the urinary tract
* SGPT < 2.5 times normal
* Bilirubin < 1.5 mg/dL
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by MUGA
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study and for ≥ 1 month after study completion
* No evidence of uncontrolled infection
* Able to undergo radiotherapy NOTE: *Abnormal blood counts allowed if there is bone marrow biopsy or aspirate proven bone marrow involvement by rhabdomyosarcoma

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy except steroids
* No prior radiotherapy
* No concurrent aprepitant during ifosfamide or doxorubicin hydrochloride chemotherapy
* No concurrent dexrazoxane
* No concurrent sargramostim (GM-CSF) or pegfilgrastim

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2006-07; Primary Completion 2010-01 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Weigel, MD, Study Chair — Masonic Cancer Center, University of Minnesota; Carola A Arndt, MD, Study Chair — Mayo Clinic
Locations (166):
- United States (143):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - University of Illinois Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - Saint Louis, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - John Hunter Hospital, Newcastle, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital, Herston, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Swiss Pediatric Oncology Group Bern, Bern, Switzerland

REFERENCES:
- [Result] Weigel B, Lyden E, Anderson JR, et al.: Early results from Children's Oncology Group (COG) ARST0431: intensive multidrug therapy for patients with metastatic rhabdomyosarcoma (RMS). [Abstract] J Clin Oncol 28 (Suppl 15): A-9503, 2010.
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- High_Risk_Rhabdomyosarcoma: Parameningeal (without intracranial extension) and paraspinal tumors receive chemotherapy starting Week 1 and begin radiation therapy at Week 20. Weeks 1-6: vincristine sulfate and irinotecan hydrochloride. Weeks 7-34: vincristine sulfate and irinotecan hydrochloride, Cyclophosphamide with MESNA, Doxorubicin hydrochloride, Etoposide, Ifosfamide with MESNA. Weeks 35-54: vincristine sulfate, Dactinomycin, irinotecan hydrochloride and Cyclophosphamide with MESNA and Filgrastim. Radiation therapy beginning at Week 20. Second look conventional surgery: Surgical resection other than biopsy will be applicable for the majority of patients.
Period: Overall Study
Arm/Group | High_Risk_Rhabdomyosarcoma
Started | 109
Completed | 67
Not Completed | 42
Not completed — Adverse Event | 2
Not completed — Death | 2
Not completed — Lack of Efficacy | 11
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 11
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Arm/Group | High_Risk_Rhabdomyosarcoma
Number analyzed (Participants) | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 96
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.85 (6.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 76
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 92
  Canada | 11
  Australia | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete or Partial Response Assessed by RECIST Criteria
Description: Volumetric measurements of the primary tumor using an elliptical model (0.5 x the product of the 3 largest perpendicular diameters) to assess response to neoadjuvant therapy. The RECIST (Response Evaluation Criteria in Solid Tumors) from the NCI will be used for assessment of the size of measurable metastases, including nodal metastases. Primary Tumor Measurement: Technical guidelines for cross-sectional imaging computed tomography (CT) slice thickness should be 5mm or less and the diameter of the "measurable" mass should be at least twice the reconstructed slice thickness. Smaller masses are considered detectable, but will be counted as "non-measurable." Complete Response (CR): Complete disappearance of the tumor confirmed at >4 weeks. Partial Response (PR): At least 64% decrease in volume compared to the measurement obtained at study enrollment. Progressive Disease (PD): At least 40% increase in tumor volume compared to the smallest volume obtained since the beginning.
Time Frame: Protocol week 6 evaluation
Population: All eligible patients with protocol week tumor assessment (N=102)
Measure: Number; unit: percentage of participants
Arm/Group | High_Risk_Rhabdomyosarcoma
Number analyzed (Participants) | 102
percentage of participants | 63

2. Primary Outcome: Percentage of Patients Experiencing Adverse Events Due to Concurrent Therapy
Description: Adverse events are reported for patients receiving concurrent irinotecan hydrochloride and radiotherapy.
Time Frame: From enrollment to up to 2 years
Population: Percentage of patients experiencing a grade 3/4/5 toxicity in a course.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | High_Risk_Rhabdomyosarcoma
Number analyzed (Participants) | 109
percentage of patients
  Course 1 | 53.3 [43.4 to 63.0]
  Course 2 | 68.4 [58.2 to 77.4]
  Course 3 | 79.3 [69.3 to 87.3]
  Course 4 | 55.7 [43.3 to 67.6]

3. Secondary Outcome: Percentage of Patients Event Free at 4 Years Following Study Entry
Description: Event-free survival: Time to recurrence, second malignancy, or death as a first event, estimated from a Kaplan Meier curve
Time Frame: 4 years
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- High_Risk_Rhabdomyosarcoma: Patients with parameningeal (without intracranial extension) and paraspinal tumors should receive chemotherapy beginning Week 1 and begin radiation therapy at Week 20. Weeks 1-6 vincristine sulfate (VCR) & irinotecan hydrochloride (IRIN), Weeks 7-34 vincristine sulfate (VCR), Cyclophosphamide (CPM) with MESNA, Doxorubicin hydrochloride (DOX), Etoposide (ETOP), Ifosfamide (IFOS) with MESNA. Weeks 35-54 vincristine sulfate (VCR), Dactinomycin (DACT) and Cyclophosphamide (CPM) with MESNA and Filgrastim. Radiation therapy beginning at Week 20. Second look conventional surgery: Surgical resection other than biopsy will be applicable for the majority of patients.
Arm/Group | High_Risk_Rhabdomyosarcoma
Number analyzed (Participants) | 109
Percentage of patients | 36 [27 to 46]

ADVERSE EVENTS:
Description: The denominator for adverse events is 108 rather than 109 is because 1 patient did not receive treatment, therefore was excluded from the denominator.
Arm/Group | High_Risk_Rhabdomyosarcoma
Serious Adverse Events (participants affected / at risk) | 4/108
Other Adverse Events (participants affected / at risk) | 95/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High_Risk_Rhabdomyosarcoma (N=108)
Anorectal infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High_Risk_Rhabdomyosarcoma (N=108)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal infection (Infections and infestations) | 2
Abdominal pain (Gastrointestinal disorders) | 15
Acidosis (Metabolism and nutrition disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 12
Alkalosis (Metabolism and nutrition disorders) | 1
Anal pain (Gastrointestinal disorders) | 3
Anaphylaxis (Immune system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 8
Anorectal infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 24
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bladder infection (Infections and infestations) | 3
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Blood antidiuretic hormone abnormal (Investigations) | 1
Blood bilirubin increased (Investigations) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac disorders - other (Cardiac disorders) | 1
Catheter related infection (Infections and infestations) | 8
Chronic kidney disease (Renal and urinary disorders) | 1
Cognitive disturbance (Nervous system disorders) | 2
Colitis (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 2
Cystitis noninfective (Renal and urinary disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 17
Depression (Psychiatric disorders) | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 6
Diarrhea (Gastrointestinal disorders) | 34
Dysphagia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Enterocolitis infectious (Infections and infestations) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Esophageal pain (Gastrointestinal disorders) | 2
Esophageal stenosis (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 44
Fever (General disorders) | 4
Gait disturbance (General disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2
General disorders and administration site conditions - Other (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
GGT increased (Investigations) | 3
Headache (Nervous system disorders) | 5
Hematuria (Renal and urinary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 20
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypotension (Vascular disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Ileus (Gastrointestinal disorders) | 3
Infections and infestations - Other (Infections and infestations) | 51
INR increased (Investigations) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Lipase increased (Investigations) | 4
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
Malabsorption (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 20
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nail infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 21
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 9
Non-cardiac chest pain (General disorders) | 2
Oral pain (Gastrointestinal disorders) | 4
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pain (General disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 8
Peripheral nerve infection (Infections and infestations) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8
Personality change (Psychiatric disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Platelet count decreased (Investigations) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural infection (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Proctitis (Gastrointestinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rectal mucositis (Gastrointestinal disorders) | 2
Rectal pain (Gastrointestinal disorders) | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Serum amylase increased (Investigations) | 1
Sinus pain (Nervous system disorders) | 1
Skin infection (Infections and infestations) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Tooth infection (Infections and infestations) | 1
Typhlitis (Gastrointestinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Vascular disorders - Other (Vascular disorders) | 1
Venous injury (Injury, poisoning and procedural complications) | 1
Vomiting (Gastrointestinal disorders) | 16
Weight loss (Investigations) | 14
White blood cell decreased (Investigations) | 4
Wound infection (Infections and infestations) | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No